CLINICAL TRIAL: NCT00176072
Title: B l u e C Q - P r o j e c t: Bioavailability of Methylene Blue (MB) - Comparison of an Intravenous and Two Oral Formulations - and Influence of Sustained Release MB on Chloroquine (CQ) Concentrations
Brief Title: BlueCQ Bioavailability
Status: Completed | Type: Observational
Sponsor: Heidelberg University (Other)
Other Study IDs: K102
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2004-07

CONDITIONS: Methylene Blue; Chloroquine; Pharmacokinetics; Bioavailability

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
Bioavailability of methylene blue (MB) - comparison of an i.v. and two oral MB formulations - and influence of sustained release MB on chloroquine (CQ) concentrations in whole blood, plasma and urine.

Intraindividual cross over open comparison in healthy male and female individuals (6:6) with different MB formulations in randomised order for the determination of the absolute bioavailability of MB (part 1), followed by an explorative randomised parallel group comparison of CQ disposition when CQ is given alone (3 males and 3 females) or in combination with 1000 mg sustained release MB (3 males and 3 females) in the participants of study part 1 (part 2).

DETAILED DESCRIPTION:
Maximum whole blood methylene blue (MB) concentrations after i.v. and oral administration may differ in the magnitude of 100:1. For achieving MB concentrations possibly effective against malaria when using different pharmaceutical formulations, determination of oral bioavailability of MB is necessary. To investigate this 12 healthy subjects (6 females, 6 males) will receive in a randomised cross over design MB 50 mg i.v. and MB 500 mg as a oral solution.

For generating this information for a planned phase II/III study in Africa, an intravenous and an oral MB preparation will be investigated.

A second part of the study will explorative investigate the influence of MB on chloroquine (CQ) plasma concentrations. During this part 6 healthy subjects (3 females, 6 males) will receive either CQ alone or in combination with MB 500 mg, the design of this part will be a parallel design.

ELIGIBILITY:
Inclusion Criteria:

Good state of health physically and mentally

Exclusion Criteria:

Any regular drug treatment currently or past (within the last 2 months) except for oral contraceptives in females Treatment with a known inhibitor or inducer of drug metabolising enzymes or transport proteins within a period of less than 10 times the respective elimination half-life

Any acute or chronic illness, especially:

Glucose-6-phosphate dehydrogenase deficiency Allergic disposition or history of hypersensitivity reactions Smoking Alcohol or drug abuse

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18
Dates: Start 2004-08; Study Completion 2004-11

CONTACTS AND LOCATIONS:
Overall Officials: Gerd Mikus, MD Bsc, Principal Investigator — Department Internal Medicine VI